CLINICAL TRIAL: NCT00677287
Title: Phase I/II Study of Multiple-Vaccine Therapy Using Epitope Peptide Restricted to HLA-A*2402 in Combination With Tegafur/Uracil/Folinate in Treating Patients With Refractory Colorectal Cancer
Brief Title: Histocompatibility Leukocyte Antigen (HLA)-A*2402 Restricted Peptide Vaccine Therapy in Patients With Colorectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of financial support
Sponsor: Tokyo University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Department of Surgery, The Institute of Medical Science, The University of Tokyo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC-A24-I, II
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2008-05

CONDITIONS: Colorectal Cancer; Colon Cancer; Rectal Cancer
Keywords: HLA-A*2402; Peptide Vaccine; RNF43; TOMM34; VEGFR1; VEGFR2
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — RNF43 protein, human; Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Biological: RNF43, TOMM34, VEGFR1 and VEGFR2

INTERVENTIONS:
Biological: RNF43, TOMM34, VEGFR1 and VEGFR2 — Patients will be vaccinated twice a week for 8 weeks. On each vaccination day, RNF43 peptide (1mg), TOMM34 peptide (1mg), VEGFR1 peptide (1mg) and VEGFR2 peptide (1mg) mixed with Montanide ISA 51 will be administered by subcutaneous injection in combination with Tegafur/Uracil/Folinate chemotherapy.

SUMMARY:
The purpose of this study is to evaluate the safety and time to progression of HLA-A*2402 restricted epitope peptides RNF43, TOMM34, VEGFR1 and VEGFR2 emulsified with Montanide ISA 51 in combination with Tegafur/Uracil/Folinate chemotherapy.

DETAILED DESCRIPTION:
RNF43 and TOMM34 have been identified as cancer specific molecules especially in colorectal cancer using genome-wide expression profile analysis by cDNA microarray technique. VEGF receptor 1 and 2 are essential targets to tumor angiogenesis, and we identified that peptides derived from these receptors significantly induce the effective tumor specific CTL response in vitro and vivo. According to these findings, in this trial, we evaluate the safety, immunological and clinical response of those peptides. Patients will be vaccinated twice a week for 8 weeks. On each vaccination day, RNF43 peptide (1mg), TOMM34 peptide (1mg), VEGFR1 peptide (1mg) and VEGFR2 peptide (1mg) mixed with Montanide ISA 51 will be administered by subcutaneous injection. The patients will also receive oral chemotherapy (Tegafur/Uracil/Folinate) simultaneously. Repeated cycles of the vaccine and the chemotherapy will be administered until patients develop progressive disease or unacceptable toxicity, whichever occurs first. In the phase I study, we evaluate the safety and tolerability of these peptide vaccine. In the following phase II study, we evaluate the immunological and clinical response of this vaccine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or recurrent colorectal cancer
* Resistant against chemotherapy including CPT-11, l-OHP、+/- 5-FU +/- bevacizumab or difficult to continue the chemotherapy due to intolerable side effect(s)
* ECOG performance status 0-2
* Life expectancy > 3 months
* HLA-A*2402
* Laboratory values as follows

  * 2000/mm3<WBC<15000/mm3
  * Platelet count>100000/mm3
  * Bilirubin < 3.0mg/dl
  * Asparate transaminase < 150IU/L
  * Alanine transaminase < 150IU/L
  * Creatinine < 3.0mg/dl
* Able to receive oral Tegafur/Uracil/Folinate therapy
* Able and willing to give valid written informed consent

Exclusion Criteria:

* Pregnancy(woman of childbearing potential:Refusal or inability to use effective means of contraception)
* Breastfeeding
* Active or uncontrolled infection
* Unhealed external wound
* Concurrent treatment with steroids or immunosuppressing agent
* Prior chemotherapy,radiation therapy, or immunotherapy within 4 weeks
* Uncontrolled brain and/or intraspinal lesion(s)
* History of allergy to Tegafur, Uracil, and/or Folinate
* Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
safety(Phase I:toxicities as assessed by NCI CTCAE version3) and efficacy(Phase II:Feasibility as evaluated by RECIST) | 2 months

SECONDARY OUTCOMES:
To evaluate immunological responses | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Masaru Shinozaki, MD/PhD, Principal Investigator — Head, Department of Surgery
Locations (1):
- The Institute of Medical Science, the University of Tokyo, Minato-ku, Tokyo, Japan

REFERENCES:
- [Background] Uchida N, Tsunoda T, Wada S, Furukawa Y, Nakamura Y, Tahara H. Ring finger protein 43 as a new target for cancer immunotherapy. Clin Cancer Res. 2004 Dec 15;10(24):8577-86. doi: 10.1158/1078-0432.CCR-04-0104. PMID 15623641
- [Background] Shimokawa T, Matsushima S, Tsunoda T, Tahara H, Nakamura Y, Furukawa Y. Identification of TOMM34, which shows elevated expression in the majority of human colon cancers, as a novel drug target. Int J Oncol. 2006 Aug;29(2):381-6. PMID 16820880
- [Background] Niethammer AG, Xiang R, Becker JC, Wodrich H, Pertl U, Karsten G, Eliceiri BP, Reisfeld RA. A DNA vaccine against VEGF receptor 2 prevents effective angiogenesis and inhibits tumor growth. Nat Med. 2002 Dec;8(12):1369-75. doi: 10.1038/nm1202-794. Epub 2002 Nov 4. PMID 12415261
- [Background] Li Y, Wang MN, Li H, King KD, Bassi R, Sun H, Santiago A, Hooper AT, Bohlen P, Hicklin DJ. Active immunization against the vascular endothelial growth factor receptor flk1 inhibits tumor angiogenesis and metastasis. J Exp Med. 2002 Jun 17;195(12):1575-84. doi: 10.1084/jem.20020072. PMID 12070285
- [Background] Ishizaki H, Tsunoda T, Wada S, Yamauchi M, Shibuya M, Tahara H. Inhibition of tumor growth with antiangiogenic cancer vaccine using epitope peptides derived from human vascular endothelial growth factor receptor 1. Clin Cancer Res. 2006 Oct 1;12(19):5841-9. doi: 10.1158/1078-0432.CCR-06-0750. PMID 17020992
- [Background] Wada S, Tsunoda T, Baba T, Primus FJ, Kuwano H, Shibuya M, Tahara H. Rationale for antiangiogenic cancer therapy with vaccination using epitope peptides derived from human vascular endothelial growth factor receptor 2. Cancer Res. 2005 Jun 1;65(11):4939-46. doi: 10.1158/0008-5472.CAN-04-3759. PMID 15930316
- See also: Research Hospital, the Institute of Medical Science, the University of Tokyo — http://www.transrec.jp/